CLINICAL TRIAL: NCT02465827
Title: Selective Blocks for Total Knee Arthroplasty
Brief Title: Ultrasound-guided Selective Blockade of the Saphenous and Obturator Nerves Following Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Jens Borglum Neimann, Ass professor, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BispebjergH
Record Dates: First submitted 2015-06-02; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Knee Arthroplasty, Total
MeSH Terms: interventions — Nerve Block; Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saphenous and obturator nerve block (Active Comparator): 5 ml of ropivacaine 0.75% for the saphenous nerve and 10 ml of ropivacaine 0,75% for the obturator nerve block.
  Ropivacaine 0.75% for nerve blockades for both nerves mentioned.
  Interventions: Drug: nerve block with ropivacaine
- Saphenous nerve block (Active Comparator): 5 ml of ropivacaine 0.75% for the saphenous nerve and 10 ml of isotonic saline for the obturator nerve block.
  Ropivacaine 0.75% for the saphenous nerve block and saline for the obturator nerve block
  Interventions: Drug: nerve block with ropivacaine and with saline
- Placebo nerve block (Placebo Comparator): 5 ml of isotonic saline for the saphenous nerve and 10 ml of isotonic saline for the obturator nerve block.
  Saline for nerve blockades for both nerves mentioned.
  Interventions: Drug: nerve block with saline

INTERVENTIONS:
Drug: nerve block with ropivacaine — Ultrasound guided nerve blocks of the saphenous and obturator nerve, posterior branch with ropivacaine 0.75% for both nerve branches
  Other Names: Saphenous and obturator nerve block with ropivacaine
  Arms: Saphenous and obturator nerve block
Drug: nerve block with ropivacaine and with saline — nerve blocks of the saphenous nerve with ropivacaine 0.75% and obturator nerve, posterior branch with saline
  Other Names: Saph block with ropivacaine and obtur block with saline
  Arms: Saphenous nerve block
Drug: nerve block with saline — Ultrasound guided nerve blocks of the saphenous and obturator nerve, posterior branch with saline for both nerve branches
  Other Names: saphenous and obturator nerve block with saline
  Arms: Placebo nerve block

SUMMARY:
The investigators aimed to evaluate the efficacy of selective low volume ultrasound-guided blockades of the saphenous and obturator nerves on dynamic and rest pain 24-hours post-operatively for patients undergoing unilateral primary total knee arthroplasty.

DETAILED DESCRIPTION:
A femoral nerve block is the recommended strategy in many surgical centers to supplement multimodal analgesic regime following total knee arthroplasty (TKA) (i.e. both for spinal and general anesthesia). However, a femoral nerve block will often result in quadriceps paralysis, and this will increase the risk for the patient to fall as long as the femoral block have effect. Thus, the search for sensory nerve blocks to stop pain after TKA is a very interesting topic. The saphenous nerve is a purely sensory nerve, and the posterior branch of the obturator nerve is a mixed nerve, where the motor component only affects part of the adductor major muscle.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists' physical classification I-III
2. Age ≥ 18 years undergoing primary unilateral total knee arthroplasty

Exclusion Criteria:

1. Inability to cooperate
2. Inability to speak and understand Danish
3. Allergy to any drugs used in the study
4. Drug or alcohol abuse
5. Pregnancy or nursing
6. Opioid abusers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Dynamic pain (pain upon movement) quantified as area-under-the-curve (AUC) 24-hours post-operatively | 24 hours
  NRS 0-10

SECONDARY OUTCOMES:
Pain at rest quantified as area-under-the-curve (AUC) 24-hours post-operatively | 24 hours
  NRS 0-10
Total opioid consumption | 24 hours
  mg
Nausea and vomiting | 24 hours
  NRS 0-10
Time to first mobilization | 24 hours
  hours
Length of stay in recovery and hospital | 72 hours
  hours
Number of clinical complications | 72 hours
  total number